CLINICAL TRIAL: NCT07238426
Title: ATTRACT-52: Advancing TTR Testing and Risk-Based Amyloidosis Cardiac Screening in Primary Care - The Ordu Pilot Study
Brief Title: ATTRACT-52: Primary Care Cardiac Amyloidosis Screening in Ordu, Turkey
Acronym: ATTRACT-52
Status: Not yet recruiting | Type: Observational
Sponsor: Kotyora Family Medicine Health Management and Education Association (Network)
Collaborators: Ordu University, Faculty of Medicine - Department of Cardiology (Academic Collaborator) (Unknown); Ordu Provincial Health Directorate - Family Medicine Network (Regional Collaborator) (Unknown)
Responsible Party: Sponsor
Other Study IDs: KAHSED-001; KAHSED-001 (Other: Kotyora Family Medicine Health Management and Education Association (KAHSED)); pending (Other: Ordu University Non-Interventional Clinical Research Ethics Committee)
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Amyloidosis; Transthyretin Amyloidosis
Keywords: ATTR-CM; primary care; family medicine; NT-proBNP; HFpEF
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Risk-based Screening Cohort: Adults ≥65 years in primary care screened using predefined red flags; high-suspicion cases receive NT-proBNP/BNP testing before referral per standard care.

SUMMARY:
Cardiac amyloidosis is a progressive infiltrative cardiomyopathy, most commonly related to transthyretin (ATTR) misfolding. Although considered rare, emerging data suggest higher prevalence in specific regions, including the Black Sea area of Turkey. Early recognition improves outcomes. ATTRACT-52 is a prospective, observational, non-interventional screening study in primary care (family medicine centers) across Ordu province. Adults ≥65 years with cardiac or musculoskeletal "red flags" will be screened; those meeting high-suspicion criteria will undergo NT-proBNP/BNP testing at the primary care level to aid risk stratification prior to referral for confirmatory diagnostics.

DETAILED DESCRIPTION:
This study implements a risk-based screening pathway for suspected transthyretin cardiac amyloidosis (ATTR-CM) in primary care. Eligible adults (≥65 years) with relevant cardiac diagnoses (e.g., heart failure, aortic stenosis, cardiomyopathy, AV block, atrial fibrillation) and/or extracardiac red flags (e.g., carpal tunnel syndrome, spinal stenosis, trigger finger) will be reviewed against predefined criteria. When high suspicion is present, NT-proBNP (>600 pg/mL) or BNP (>150 pg/mL) will be obtained in primary care to refine risk prior to referral for confirmatory testing (e.g., bone scintigraphy, CMR) per standard care. Only high-risk patients will be tested; the number of tests will remain limited and appropriate for feasibility. Primary outcomes focus on diagnostic yield and feasibility of this first-line screening model in family medicine settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Registered patient in participating Family Medicine Centers (Ordu province)
* Cardiac history including at least one of: heart failure (I50), aortic stenosis (I35.0), cardiomyopathy (I42), atrioventricular block (I44), or atrial fibrillation (I48)
* Echocardiographic interventricular septal thickness ≥12 mm with preserved LVEF (≥50%), when available
* Ability to provide verbal or written consent

Exclusion Criteria:

* Known systemic AL amyloidosis
* Severe renal impairment (eGFR <30 mL/min/1.73m²)
* Inability to provide consent
* Concurrent participation in an interventional trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged ≥65 years receiving care at Family Medicine Centers in Ordu province with cardiac and/or extracardiac red flags suggestive of possible ATTR-CM.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of high-suspicion participants with elevated NT-proBNP (>600 pg/mL) | Baseline (Day 0)
  Percentage of high-suspicion cases exceeding the predefined NT-proBNP threshold at baseline.

SECONDARY OUTCOMES:
Confirmed cardiac amyloidosis diagnosis rate | Up to 12 months
  Number and proportion of referred participants with confirmed ATTR-CM by standard diagnostics.
Time from screening to confirmed diagnosis | Up to 12 months
  Interval (days) between initial screening and definitive diagnostic confirmation.
Feasibility and physician protocol adherence | Up to 12 months
  Proportion of participating primary care physicians completing all required screening steps.

CONTACTS AND LOCATIONS:
Overall Officials: Seçkin Dereli, MD, Assoc. Prof., Principal Investigator — Ordu University Faculty of Medicine, Department of Cardiology (Turkey)

IPD SHARING:
Plan to Share IPD: No
Not planned for this pilot observational screening study.